CLINICAL TRIAL: NCT00087867
Title: An Open-label Study of the Efficacy, Safety, and Tolerability of Oral SCIO-469 in Treatment of Relapsed, Refractory Patients With Multiple Myeloma
Brief Title: Study of Oral SCIO-469 in Relapsed, Refractory Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Responsible Party: VP Clinical Oncology, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005152; SCIO-469MMY2001 (B003)
Record Dates: First submitted 2004-07-14; First posted 2004-07-19 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; SCIO-469; p38 MAP kinase; myeloma; bone marrow
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — SCIO-469; Bortezomib

ARMS (2):
- 001 (Experimental): SCIO-469 two 30-mg capsules three times daily
  Interventions: Drug: SCIO-469
- 002 (Other): SCIO-469 and bortezomib In addition to SCIO-469 patients with disease progression will receive bortesomib 1.0 mg/m2 intravenously as a bolus injection on Days 1 4 8 and 11 of a 21-day cycle followed by a 10-day rest period
  Interventions: Drug: SCIO-469 and bortezomib

INTERVENTIONS:
Drug: SCIO-469 — two 30-mg capsules three times daily
  Arms: 001
Drug: SCIO-469 and bortezomib — In addition to SCIO-469, patients with disease progression will receive bortesomib 1.0 mg/m2 intravenously as a bolus injection on Days 1, 4, 8, and 11 of a 21-day cycle, followed by a 10-day rest period
  Arms: 002

SUMMARY:
The main objective of this study is to assess the efficacy of SCIOS-469 as monotherapy in relapsed, refractory patients with multiple myeloma (MM), based on response rates.

DETAILED DESCRIPTION:
The main objective of this study is to assess the efficacy of SCIO-469 as monotherapy in relapsed, refractory patients with multiple myeloma (MM), based on response rates. Patients took SCIO-469 two capsules (60 mg) by mouth three times a day with water, preferably with a meal, for 72 days except on Days 1 and 30 of monotherapy and Days 1 and 11 of combination therapy. On these days, the second dose of SCIO-469 was administered after collection of the 12-hour PK sample, and the third dose was not administered.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy more than three months
* diagnosed with multiple myeloma (MM)
* relapsed following a response to any conventional MM therapy, and refractory to their most recent MM therapy
* Karnofsky performance status = 60
* no electrocardiographic evidence of acute ischemia or new conduction system abnormalities
* no history of myocardial infarction within last 6 months
* serum concentrations of aspartate aminotransferase (AST) and alanine aminotransferase (ALT) = 3X upper limit of normal (ULN)
* total serum bilirubin = 2X ULN
* Calculated or measured creatinine clearance >30 mL/min
* platelet count = 30 x 10(9)/L
* hemoglobin concentration = 8 g/dL
* white blood cell count = 2.0 x 10(9)/L

Exclusion Criteria:

* Patients with non-secretory myeloma, plasma cell leukemia, or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, M-protein and skin changes)
* major surgery within four weeks of enrollment
* severe elevated serum calcium
* heart failure
* receipt of chemotherapy within 21 days before enrollment, receiving immunotherapy, radiation therapy, or other investigational agents
* receipt of corticosteroids equivalent to more than 10 mg/day of prednisone within two weeks before enrollment
* known allergies to agents used in bortezomib (e.g., boron or mannitol)
* poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-06; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Patient responses (CR, PR, MR, and overall response) are assessed using EBMT criteria, which primarily involve assessments of monoclonal paraprotein in the serum and urine and assessment of changes in soft tissue plasmacytomas and bone lesions. | Day 73

SECONDARY OUTCOMES:
Time to first response, time to best response, and percentage of patients with disease progression were assessed. | Days 1, 15, 30, 52, and 73
Size and number of lytic bone lesions were summarized. | screening and Day 73
Quality of life and pain was assessed. | Days 1, 15,30,52,73
Performance status was evaluated. | Screening, Days 1, 30, 73
Bone disease was monitored by assessing various markers. | Days 1, 15, 30, 52, 73

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.